CLINICAL TRIAL: NCT03733080
Title: Large-scale Online Studies of Motor Responses and Cognition
Brief Title: Large-Scale Online Studies of Early Motor Skill Learning
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999919012; 19-N-N012
Record Dates: First submitted 2018-11-06; First posted 2018-11-07 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Healthy
Keywords: AMT; Natural History

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: ages 18 and older

SUMMARY:
Background:

Our goal is to gain insight into early human motor skill learning by carrying out online substudies using online crowd-sourcing tools.

Objective:

To learn more about motor behavior in a large group of people using motor tasks, and questions.

Eligibility:

Adults ages 18 and older based in the U.S. who speak English

Design:

Participants will be recruited from a crowd-sourcing website like Amazon Mechanical Turk.

Participants will do online tasks. They can use their own computers anywhere with Internet access. They will not need to directly interact with researchers.

Participants will be asked for general data, like their age and gender. No personally identifiable data will be collected.

Participants will see a list of tasks on their computer screen. They will be able to choose tasks they wish to do. They will get a description of the experiment, how long it takes, and how much compensation they will get.

Participants will complete on their screen a motor behavioral task, a cognitive task, and/or a questionnaire. For example, they may be asked to press sequences of numbers on the keyboard or move the mouse when a stimulus appears on the screen. Experiments may last up to 1 hour.

Participants can complete as many experiments as they wish. They can quit at any point.

DETAILED DESCRIPTION:
Objective:

Our overall goal in this protocol has been to gain insight into early motor skill learning (micro-learning) in large-scale healthy volunteer cohorts using online crowd-sourcing. We have used a simple keyboard typing task to study micro-offline performance improvements during early motor skill learning. This online approach limits the burden on participants (who perform tasks in the comfort of their homes instead of traveling to NIH) and substantially reduces burden on in-house human, financial and technical resources. Results from this protocol contribute to a better understanding of factors relevant to human motor skill learning, with important implications for the design of better motor learning and neurorehabilitative strategies after brain lesions. We had completed data collection for four aims under this protocol at the time we were informed by the NIH IRB that they determined this to be a thematic protocol (September 23, 2019).

The four specific aims addressed under this protocol are:

1. Aim 1. To validate a motor skill learning task previously used by our group in lab-based studies {Bonstrup, 2019 #36} within an online, crowd-sourcing platform.
2. Aim 2. To compare the influence of an interfering task applied during early ("early interference") vs late ("late interference") rest periods on motor learning, thus evaluating resistance to interference, a feature of consolidation.
3. Aim 3. To evaluate the effects of a shorter practice period duration (i.e. - 5s vs. previously studied 10s duration) on micro-offline motor learning to gain insight into the impact of fatigue-related factors on learning.
4. Aim 4. To evaluate the effects of randomly variable practice period durations between 5-10s in length on micro-offline gains

As instructed, the purpose of this amendment is to request authorization to proceed with data analysis and publication. No new experiments will be carried out under this protocol.

Study Population:

U.S.-based English speakers aged 18 and above were recruited under this minimal risk protocol. Participants completed an online task in the comfort of their own homes using the internet, and did not need to directly interact with the investigators. All participants were given an anonymized random ID by the on-line site. We did collect general demographic information including age (needed to determine elegibility), and gender, race and ethnicity (per IRB reporting requirements, i.e. - Cumulative Inclusion Enrollment Report). However, we did not collect personally identifiable information (PII) about the participants.

Design:

Under this protocol, we have conducted experiments supporting four aims using Amazon Mechanical Turk (AMT). All experiments consisted of a brief keyboard typing task where participants were asked to repeatedly type a 5-key sequence (4-1-3-2-4) as fast and as accurately as possible for several seconds (i.e. - practice trial). Each practice trial was followed by a rest period lasting several seconds. Following the task, participants completed a short questionnaire designed to query compliance with task instructions, and collect general demographic data required for IRB reporting. The average total time for participation across all experiments was approximately 20 minutes.

Outcome Measures:

The primary outcome measures for the keyboard typing task were correct sequence typing speed and typing accuracy. Microlearning scores were derived by quantifying the speed change between the end of a previous practice trial and the beginning of the subsequent one (micro-offline learning) and the speed difference between the beginning and end of the same practice trial (micro-online learning). Information from the questionaires related to task instruction compliance was primarily used to exclude data from further analysis if needed.

ELIGIBILITY:
* INCLUSION CRITERIA:

U.S.-based English speakers greater than 18 years of age are eligible to participate in the study.

EXCLUSION CRITERIA:

Subjects are excluded if they are less than 18 years of age. NIH and NINDS employees are not excluded from the study, since participation is anonymous and personal identifiers unknown to the experimenters.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 2,529 volunteers have participated in this protocol. It is possible that some of these participants may have been NIH or NINDS employees, since participant identities were anonymous to the experimenters. Data aquired from 97 participants was used for testing and debugging the typing task application during initial technical development. These data are not useable for research purposes.
Sampling Method: Probability Sample
Enrollment: 2529 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2019-10-17 (Actual); Study Completion 2019-10-17 (Actual)

PRIMARY OUTCOMES:
data analysis | in data analysis
  Aim 1. To validate a motor skill learning task previously used by our group in lab-based studies {Bonstrup, 2019 #36} within an online, crowd-sourcing platform. Aim 2. To compare the influence of an interfering task applied during early ( early interference group) vs late ( late interference ) rest periods on stabilization of motor learning. Aim 3. To evaluate the effects of shorter practice period durations (i.e. - 5s vs. previously studied 10s duration) on micro-offline motor learning to gain insight into the impact of fatigue-relatedfactors on learning. Aim 4. To evaluate the effects of randomly variable practice period durations between 5-10s in length on micro-offline gains

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo G Cohen, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States